CLINICAL TRIAL: NCT00960414
Title: Supporting Health by Integrating Nutrition and Exercise (SHINE)
Brief Title: Randomized Controlled Clinical Trial of Weight Loss Programs in Obese Persons
Acronym: SHINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P01AT005013 (NIH); P01AT005013 (NIH)
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Results first posted 2024-02-14 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Obesity
Keywords: obesity; randomized controlled trial; weight loss; metabolic syndrome
MeSH Terms: conditions — Obesity; Weight Loss; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SHINE A (Experimental): Mindfulness training added to diet-exercise education.
  Interventions: Behavioral: SHINE
- SHINE B (Active Comparator): Diet-exercise education.
  Interventions: Behavioral: SHINE

INTERVENTIONS:
Behavioral: SHINE — Both groups will receive a diet and exercise based intervention aimed at eating a caloric intake that will maintain ideal body weight and increasing exercise. SHINE A will emphasize awareness of hunger and satiety cues, while SHINE B will receive more detailed nutritional education.

SUMMARY:
The purpose of this study is to compare two approaches to a diet and exercise-based weight loss program.

DETAILED DESCRIPTION:
The high prevalence of obesity and its medical consequences make it one of the most important public health issues in the United States today. Few interventions have been consistently successful at reducing obesity. This trial will test an intervention program that lasts 22 weeks, with 16 evening sessions and one weekend day. Participants will be randomized to one of two arms. Both arms will receive diet and exercise intervention elements. The study aims for gradual weight loss, with a calorie target that will maintain ideal body weight, rather than a more calorie restricted diet. The exercise component is based around increasing walking. The arms will compare methods for producing long-lasting behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years old
* BMI > 30-45
* Waist circumference > 102 cm (men) or > 88 cm (women)
* Live in San Francisco Bay Area and able to attend more than 16 classes and up to 12 assessment visits in San Francisco over an 18 month period

Exclusion Criteria:

* Inability to provide informed consent
* Age < 18
* A substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate in the group intervention
* Type I or II Diabetes or fasting glucose ≥ 126 mg/dl or hemoglobin A1c ≥ 6.5; those with HbA1c between 6-6.5% may complete an OGTT to rule out diabetes (glucose <200 mg/dl)
* Use of systemic (oral or IV) corticosteroids in the 6 months prior to enrollment or severe autoimmune disorders or other conditions (e.g. rheumatoid arthritis, lupus), that are likely to require these medications
* Use of immunosuppressive or immunomodulating drugs or chronic or acute conditions that would require the use of such medications
* A history of known coronary artery disease (CAD), or typical or atypical anginal chest pain requires a letter from the participant's physician that he or she has been adequately evaluated and that a moderate exercise program is appropriate
* Non English speaker
* Pregnant or planning to get pregnant in the next 12 months, breastfeeding or less than 6 months post-partum
* Initiation of new class of psychiatric medications in past 2 months
* Currently on a specific weight loss diet
* For influenza vaccine administration: a prior allergic reaction to the influenza vaccine or eggs. These participants can be included in the trial but will be excluded from participation in influenza vaccination.
* Active bulimia or strong history of bulimia
* Current use of weight loss medications or supplements such as amphetamine-based drugs that are believed to have some effect on weight
* History of or planned weight loss surgery
* Untreated hypothyroidism: TSH > 4mU/mL (or the upper limit of normal reference defined by the lab doing the assay)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2009-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Hecht, MD, Principal Investigator — University of California, San Francisco; Elissa Epel, PhD, Study Chair — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Medicine, San Francisco, California, United States

REFERENCES:
- [Derived] Jake-Schoffman DE, Brown SD, Baiocchi M, Bibeau JL, Daubenmier J, Ferrara A, Galarce MN, Hartogensis W, Hecht FM, Hedderson MM, Moran PJ, Pagoto SL, Tsai AL, Waring ME, Kiernan M. Methods-Motivational Interviewing Approach for Enhanced Retention and Attendance. Am J Prev Med. 2021 Oct;61(4):606-617. doi: 10.1016/j.amepre.2021.04.005. PMID 34544560
- [Derived] Daubenmier J, Chao MT, Hartogensis W, Liu R, Moran PJ, Acree MC, Kristeller J, Epel ES, Hecht FM. Exploratory Analysis of Racial/Ethnic and Educational Differences in a Randomized Controlled Trial of a Mindfulness-Based Weight Loss Intervention. Psychosom Med. 2021 Jul-Aug 01;83(6):503-514. doi: 10.1097/PSY.0000000000000859. PMID 33214537
- [Derived] Radin RM, Epel ES, Daubenmier J, Moran P, Schleicher S, Kristeller J, Hecht FM, Mason AE. Do stress eating or compulsive eating influence metabolic health in a mindfulness-based weight loss intervention? Health Psychol. 2020 Feb;39(2):147-158. doi: 10.1037/hea0000807. Epub 2019 Nov 14. PMID 31724424
- [Derived] Mason AE, Hecht FM, Daubenmier JJ, Sbarra DA, Lin J, Moran PJ, Schleicher SG, Acree M, Prather AA, Epel ES. Weight Loss Maintenance and Cellular Aging in the Supporting Health Through Nutrition and Exercise Study. Psychosom Med. 2018 Sep;80(7):609-619. doi: 10.1097/PSY.0000000000000616. PMID 29901486
- [Derived] Hecht FM, Moskowitz JT, Moran P, Epel ES, Bacchetti P, Acree M, Kemeny ME, Mendes WB, Duncan LG, Weng H, Levy JA, Deeks SG, Folkman S. A randomized, controlled trial of mindfulness-based stress reduction in HIV infection. Brain Behav Immun. 2018 Oct;73:331-339. doi: 10.1016/j.bbi.2018.05.017. Epub 2018 May 26. PMID 29842903
- [Derived] Daubenmier J, Moran PJ, Kristeller J, Acree M, Bacchetti P, Kemeny ME, Dallman M, Lustig RH, Grunfeld C, Nixon DF, Milush JM, Goldman V, Laraia B, Laugero KD, Woodhouse L, Epel ES, Hecht FM. Effects of a mindfulness-based weight loss intervention in adults with obesity: A randomized clinical trial. Obesity (Silver Spring). 2016 Apr;24(4):794-804. doi: 10.1002/oby.21396. Epub 2016 Mar 9. PMID 26955895
- [Derived] Mason AE, Epel ES, Aschbacher K, Lustig RH, Acree M, Kristeller J, Cohn M, Dallman M, Moran PJ, Bacchetti P, Laraia B, Hecht FM, Daubenmier J. Reduced reward-driven eating accounts for the impact of a mindfulness-based diet and exercise intervention on weight loss: Data from the SHINE randomized controlled trial. Appetite. 2016 May 1;100:86-93. doi: 10.1016/j.appet.2016.02.009. Epub 2016 Feb 8. PMID 26867697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants for a weight loss study comparing two programs involving diet, exercise, and stress management from the community using fliers, newspaper advertisements, online postings, and referrals at UCSF clinics. Participants were enrolled in 6 rounds from July 2009-February 2012. Assessments were completed in October 2013.
Groups:
- SHINE A; SHINE B: SHINE: Both groups will receive a diet and exercise based intervention aimed at eating a caloric intake that will maintain ideal body weight and increasing exercise. SHINE A will emphasize awareness of hunger and satiety cues, while SHINE B will receive more detained nutritional education.
Period: Overall Study
Arm/Group | SHINE A | SHINE B
Started | 100 | 94
Completed | 81 | 67
Not Completed | 19 | 27

BASELINE CHARACTERISTICS:
Population: We randomized 194 participants to two arms (100 to group A, 94 to group B).
Groups:
- Total: Total of all reporting groups
Arm/Group | SHINE A | SHINE B | Total
Number analyzed (Participants) | 100 | 94 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.0) | 46.8 (12.4) | 47.0 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 81 | 160
  Male | 21 | 13 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  White | 65 | 50 | 115
  African American | 13 | 12 | 25
  Asian/Pacific Islander | 8 | 11 | 19
  Latina/Latino | 7 | 16 | 23
  Native American | 0 | 2 | 2
  Other | 7 | 3 | 10
Education [Number; unit: participants with bachelor's degree] | 69 | 56 | 125
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.4 (3.5) | 35.6 (3.8) | 35.47 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline to 18 Months
Description: weight loss at 18 month visit, approximately one year post-intervention completion, using attention-to-treat analyses of observed data
Time Frame: 18 months
Population: Two women in Arm B had weight-related variables censored at 18 months due to pregnancy.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | SHINE A | SHINE B
Number analyzed (Participants) | 81 | 65
kg | -5.0 (0.9) | -3.2 (1.0)

2. Secondary Outcome: Fat Distribution
Description: change in waist circumference from baseline to 18 mos
Time Frame: 0, 18 mo
Population: Two women in Arm B had weight-related variables censored at 18 months due to pregnancy.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | SHINE A | SHINE B
Number analyzed (Participants) | 81 | 65
cm | -4.8 (0.9) | -3.6 (1.0)

3. Secondary Outcome: Insulin Sensitivity
Description: change in HOMA from baseline to 18 months. HOMA-IR is a validated assessment of insulin resistance. HOMA-IR = fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
Time Frame: 18 mo
Population: 2 participants in Arm A and 1 participant in Arm B did not have the lab results needed to calculate HOMA-IR at 18 months.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SHINE A | SHINE B
Number analyzed (Participants) | 79 | 66
units on a scale | -.011 (0.23) | 0.50 (0.25)

4. Secondary Outcome: Change in Perceived Stress From Baseline to 18 Months
Description: Change in Perceived Stress Scale scores from baseline to 18 months (i.e. approximately one year post-intervention completion), using intention-to-treat. Scores range from 0-40, with higher scores indicating higher perceived stress (worse outcome).
Time Frame: 18 mo
Population: 8 participants in Arm A and 3 in Arm B did not complete this self-report survey at 18 months.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- SHINE A: Both groups received identical diet-exercise guidelines emphasizing modest calorie restriction (approx. 500 kcal/day), including decreasing calorie-dense nutrient-poor foods, substituting whole grains for simple carbohydrates, and increasing fresh fruits and vegetables, healthy oils, and proteins. The exercise component emphasized increasing daily activity and moderate intensity exercise, primarily through walking and strength training.
  In addition to the above, SHINE A received mindfulness training for stress management, eating, and exercise.
- SHINE B: Both groups received identical diet-exercise guidelines emphasizing modest calorie restriction (approx. 500 kcal/day), including decreasing calorie-dense nutrient-poor foods, substituting whole grains for simple carbohydrates, and increasing fresh fruits and vegetables, healthy oils, and proteins. The exercise component emphasized increasing daily activity and moderate intensity exercise, primarily through walking and strength training.
  In addition to the above, SHINE B received more detailed nutrition and exercise information, strength training with exercise bands, discussion of societal issues concerning weight loss, and some progressive muscle relation and cognitive-behavioral training.
Arm/Group | SHINE A | SHINE B
Number analyzed (Participants) | 73 | 64
units on a scale | -1.03 (0.57) | -0.11 (0.61)

5. Secondary Outcome: Change in Positive Emotions Subscale of the Differential Emotions Scale
Description: We used the 10-item positive emotions subscale of the Differential Emotions Scale (DES; Izard et al., 1991) to assess the extent to which a participant experienced positive emotions in the prior week. Participants responded on a five-point scale (0 = not at all, 4
  = extremely; total score possible range 0-40). We summed items to create a total score, with higher scores indicating more positive emotions.
Time Frame: 18 months
Population: 8 participants in Arm A and 3 in Arm B did not complete this self-report survey at 18 months.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | SHINE A | SHINE B
Number analyzed (Participants) | 73 | 64
score on a scale | 2.49 (0.67) | -0.21 (0.70)

6. Secondary Outcome: Stress Hormones
Time Frame: 0, 6, 12 mo
Reporting Status: Not Posted

7. Secondary Outcome: Autonomic Nervous System Function
Time Frame: 0, 3,6,12 months
Reporting Status: Not Posted

8. Secondary Outcome: Adipocyte Activity
Time Frame: 0, 6 mo
Reporting Status: Not Posted

9. Secondary Outcome: Influenza Vaccine Response
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 18 months per participant.
Arm/Group | SHINE A | SHINE B
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/94
Other Adverse Events (participants affected / at risk) | 0/100 | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No